CLINICAL TRIAL: NCT03559192
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Multi-center Study Investigating the Efficacy, Safety, Tolerability and Pharmacokinetics of JNJ-67953964 in Subjects With Major Depressive Disorder
Brief Title: A Study to Explore the Efficacy of JNJ-67953964 in the Treatment of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108487; 67953964MDD2001 (Other: Janssen Research & Development, LLC); 2019-000695-41 (EudraCT Number)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-in Period: Placebo (Placebo Comparator): Participants will receive matching placebo for the entire duration of the lead-in period.
  Interventions: Drug: Placebo
- Treatment Period: JNJ-67953964 or Placebo (Experimental): Participants who respond or do not respond (based on reduction from lead-in baseline in MADRS) in the placebo lead-in period will receive either matching placebo or 10 (2*5) milligram (mg) JNJ-67953964 capsules in a 1:1 ratio for 6 weeks.
  Interventions: Drug: JNJ-67953964; Drug: Placebo
- Withdrawal Period: Placebo (Placebo Comparator): Participants who complete the double-blind treatment period prior to the end of Week 11 will receive matching placebo for the remaining time of the treatment phase of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-67953964 — JNJ-67953964 10 mg will be administered as two 5-mg capsules orally once daily.
  Arms: Treatment Period: JNJ-67953964 or Placebo
Drug: Placebo — Matching placebo will be administered as 2 capsules orally once daily.

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-67953964 compared to placebo when administered as adjunctive treatment in participants with Major Depressive Disorder (MDD) partially responsive to selective serotonin reuptake inhibitor/ serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) treatment in terms of reduction of symptoms of depression, as assessed by the change from baseline on the Montgomery Asberg Depression Rating Scale (MADRS) in non-responders during the placebo lead-in period.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) between 18 and 35 kilogram per meter square (kg/m^2) inclusive (BMI = weight/height^2)
* Participants must be medically stable based on clinical laboratory tests, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and baseline
* Participants must have a primary Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) diagnosis of Major Depressive Disorder (MDD)

  1. The current episode should be less than 18 months
  2. Participants should be currently treated with an SSRI or SNRI at an adequate dose and for at least 6 weeks but no more than 12 months
  3. Have a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than or equal to (>=) 25 at screening
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before the first dose

Exclusion Criteria:

* History of documented gastric disease (including documented peptic ulcer disease, gastritis, upper gastrointestinal [GI] bleeding, esophagitis, or any GI precancerous condition), current clinically evident GI complaints
* Chronic use of a proton pump inhibitors (PPIs). History of incidental use of PPIs is allowed but should have been stopped at least 4 weeks before screening. A history of chronic nonsteroidal anti-inflammatory drug (NSAID) or aspirin use. (Low dose aspirin for example in cardiovascular disease prevention is allowed)
* Has a history of alcohol use disorder within the past year
* Has failed (no more than 25 percent [%] response on Antidepressant Treatment History Questionnaire [ATRQ]) three or more antidepressant treatments including the current Selective serotonin reuptake inhibitor/ serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) during the current depressive episode despite an adequate dose (per ATRQ) and duration (at least 6 weeks)
* Has signs or symptoms of Cushing's Disease, Addison's Disease, primary amenorrhea, or other evidence of significant medical disorders of the hypothalamus pituitary adrenal (HPA) axis
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months before the planned first dose of study drug or has participated in any interventional clinical studies on MDD in the previous 1 year or is currently enrolled in an interventional study
* Has one or more of the following diagnoses:

  1. A primary DSM (5th edition) diagnosis of generalized anxiety disorder (GAD), panic disorder, obsessive compulsive disorder (OCD), posttraumatic stress disorder (PTSD). Participants with comorbid GAD, social anxiety disorder (SAD), or panic disorder for whom MDD is considered the primary diagnosis are not excluded
  2. A current diagnosis or diagnosis in the past 1 year of psychotic disorder, MDD with psychosis, anorexia nervosa or bulimia nervosa, chronic fatigue syndrome, bipolar disorder (BD), mental retardation, antisocial or borderline personality disorder, autism spectrum disorder
* Has a current or recent history of clinically significant suicidal ideation within the past 6 months, corresponding to a score of 4 (active suicidal ideation with some intent to act, without specific plan) or 5 (active suicidal ideation with specific plan and intent) for ideation on the Colombia suicide severity rating scale (C-SSRS), or a history of suicidal behavior within the past 1 year
* Ongoing psychological treatments (example, Cognitive Behavior Therapy, Interpersonal Psychotherapy, Psychodynamic Psychotherapy, etcetera [etc.]), initiated within 1 month prior to the screening phase. A participant who has been receiving ongoing psychological treatment for a period of greater than 1 month from the screening visit is eligible, if the investigator deems the psychological treatment to be of stable duration and frequency
* Participant has a history of substance use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before screening. Mild cases can be reviewed on a case by case basis. Participants who have completed a treatment for (alcohol) addiction more than 1 year prior to first dose administration, may be included if the risk of relapse is considered minimal, total duration of alcohol use disorder was less than a year, and no significant abnormalities are shown in clinical laboratory or other pre-dose safety assessments
* Participant has used:

  1. Monoamine oxidase inhibitors (MAOIs) within 12 weeks before screening
  2. St. John's wort, ephedra, ginkgo, ginseng, or kava within 2 weeks before screening
  3. Antipsychotic drugs (D2-antagonists) within 2 weeks before screening. However, Seroquel (quetiapine) in a dose less than or equals to (<=)100 milligram (mg) is allowed when used in a stable dose for at least 8 weeks prior to screening. Quetiapine treatment should be continued unchanged during the study
  4. Opioids within 2 weeks before screening
  5. Psychostimulants such as methylphenidate or dextroamphetamine within 2 weeks before screening
  6. Psychotropics with antidepressant effects such as atomoxetine or thyroid supplementation, in addition to their SSRI or SNRI treatment within 2 weeks before screening
* Participant is unable to stop the following medication from the baseline visit (Visit 2) and throughout the study (tapering during screening period allowed): Any hypnotics including but not limited to: i. Benzodiazepines when used only as needed (PRN) are not allowed ii. Sedating antihistamines, including chronic use of diphenhydramine iii. Continuous use of zolpidem, zoplicon, eszopiclone and ramelteon. Note: Nonbenzodiazepines sleep aids (including: zolpidem, zaleplon, and eszopliclone) are allowed on an as needed (PRN) basis during the study but NOT within 24 hours before being in the clinic and not more than 2 nights in a row iv. S-adenosyl methionine (SAMe) v. Melatonin, agomelatine
* Has received any prior treatment with electroconvulsive therapy, vagal nerve stimulation, or a deep brain stimulation device or treatment with ketamine or esketamine for MDD

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (28):
  - Noble Clinical Research, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Behavioral Research Specialists LLC, Glendale, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Innova Clinical Trials, Miami, Florida
  - Galiz Research, Miami Springs, Florida
  - APG Research LLC, Orlando, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Princeton Medical Institute, Princeton, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Richmond Behavioural Associates, Staten Island, New York
  - Clinical Trials of America, Hickory, North Carolina
  - Ohio State University, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical NeuroScience Solutions Inc, Memphis, Tennessee
  - Advanced Clinical Research, West Jordan, Utah
- Germany (2):
  - Emovis GmbH, Berlin
  - Somni Bene GmbH, Schwerin
- ARENSIA, Chisinau, Moldova
- Russia (11):
  - Clinical Psychiatric Hospital #3 Named After V.A. Gilyarovsky, Moscow
  - Orenburg Regional Clinical Psychiatric Hospital #1, Orenburg
  - Medical and Rehabilitation Research Center Phoenix, Rostov-on-Don
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - City Psychiatric hospital 7 named after I.P.Pavlov, Saint Petersburg
  - Psychoneurological dispensary 1, Saint Petersburg
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Saratov Regional Psychiatric hospital named after St. Sofia, Saratov
  - Engels psychiatric hospital, Saratov Region
  - Research Institute of Mental Health, Tomsk
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg
- Ukraine (6):
  - MNCE of Kyiv RC Regional Psychiatric and Narcological Medical Association, Hlevakha
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - CNPE'Kherson Regional Institution of Mental Care'of Kherson Regional Council, Kherson
  - Cnce 'Kyiv City Psychoneurological Hospital #2' of Executive Body of Kyiv City Council (Kcsa), Kyiv
  - Mnpe 'Regional Clinical Psychiatric Hospital of Kirovohrad Regional Council', Nove
  - CNCE 'Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council', Smila
- United Kingdom (5):
  - MAC Clinical Research, Barnsley
  - MAC Clinical Research, Blackpool
  - MAC Clinical Research, Liverpool
  - Hammersmith Medicines Research Ltd, London
  - MAC Clinical Research, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Lead in Period: Placebo: Participants who successfully completed the baseline examination visit at the clinical site/unit, were treated with placebo for the entire duration of the lead-in period (up to 3 weeks).
- Double-blind Treatment + Withdrawal Period: Placebo: Participants who were responders (30 percent [%]) or more improvement on the Montgomery-Asberg Depression Rating Scale (MADRS) total score during the placebo run-in) or non-responders to lead-in placebo group were re-randomized to receive placebo matching to JNJ-67953964 capsules (2 placebo capsules) once daily during double-blind treatment period (up to 6 weeks after lead-in period) in addition to Selective serotonin reuptake inhibitors /Serotonin and norepinephrine reuptake inhibitors (SSRI/SNRI) treatment. Participants who completed the double-blind treatment period prior to the end of Week 11 entered the withdrawal period where they were treated with placebo for 2 weeks.
- Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg): Participants who were responders (30% or more improvement on the MADRS total score during the placebo run-in were responders) or non-responders to lead-in placebo group were re-randomized to receive 10 mg JNJ-67953964 capsules (2*5 mg JNJ-67953964 capsules) once daily during double-blind treatment period (up to 6 weeks after lead-in period) in addition to SSRI/SNRI treatment. Participants who completed the double-blind treatment period prior to the end of Week 11 entered the withdrawal period where they were treated with placebo for 2 weeks.
Period: Lead-in Period (3 Weeks)
Arm/Group | Lead in Period: Placebo | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Started | 181 | 0 | 0
Completed | 169 | 0 | 0
Not Completed | 12 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Period: DB Treatment(6 Wks) + Withdrawal(2 Wks)
Arm/Group | Lead in Period: Placebo | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Started | 0 | 84 | 85
Placebo Lead-in Responders | 0 | 22 | 23
Placebo Lead-In Non-Responders | 0 | 62 | 62
Completed DB Period and Entered Withdrawal | 0 | 81 | 80
Completed | 0 | 81 | 79
Not Completed | 0 | 3 | 6
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lead in Period: Placebo
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.91) [lower limit 12.91]
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 181
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 156
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 167
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Treatment Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Treatment Week 6 in Participants Who Were Non-Responders During Placebo Lead-in Period
Description: The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts. Negative change from baseline indicates improvement.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: The enriched intent-to-treat (eITT) analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
scores on a scale | -8.0 (0.92) [lower limit 0.92] | -10.1 (0.93) [lower limit 0.93]
Statistical Analysis 1: Comparison: Double-blind Treatment + Withdrawal Period: Placebo vs Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg); Test type: Superiority; p = 0.0443, Mixed Models Analysis; Least Squares Mean Difference = -2.1, 80% CI 1-sided [upper limit -1.09], Standard Error of Mean 1.25

2. Secondary Outcome: Change From Treatment Baseline in MADRS Total Score at Treatment Week 6
Description: as for outcome 1
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: The full intent-to-treat (fITT) analysis set included all enrolled participants who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-treatment baseline assessment of MADRS during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 77
scores on a scale | -6.5 (0.78) [lower limit 0.78] | -9.6 (0.79) [lower limit 0.79]
Statistical Analysis 1: Comparison: Double-blind Treatment + Withdrawal Period: Placebo vs Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg); Test type: Superiority; p = 0.0017, Mixed Models Analysis; Least Squares Mean Difference = -3.1, 80% CI 1-sided [upper limit -2.21], Standard Error of Mean 1.05

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During DB Treatment Period
Description: An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product. TEAEs were AEs with onset during the treatment period that has worsened since baseline.
Time Frame: Up to Week 6
Population: The full safety analysis set included all enrolled participants who received at least 1 dose of study medication in the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 84 | 85
Participants | 30 | 40

4. Secondary Outcome: Change From Treatment Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) Total Score at Treatment Week 6 (eITT Population)
Description: The SHAPS is a self-reported 14-item, instrument, developed for the assessment of hedonic capacity. Participants scored whether they experienced pleasure in performing a list of activities or experiences. Participants rated the answers as 1-4 where 1 indicates "Definitely agree", 2 indicates "Agree", 3 indicates "Disagree" and 4 indicates "Definitely disagree". The participant's item responses were summed to provide a total score ranging from 14 to 56. A higher total SHAPS score indicated higher levels of current anhedonia. Negative change from baseline indicated improvement.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: The eITT analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'N' (number of participants analyzed) includes the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
scores on a scale | -3.7 (0.64) [lower limit 0.64] | -4.4 (0.64) [lower limit 0.64]
Statistical Analysis 1: Comparison: Double-blind Treatment + Withdrawal Period: Placebo vs Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg); Test type: Superiority; p = 0.4188, Mixed Models Analysis; Least Squares Mean Difference = -0.7, 80% CI 1-sided [upper limit 0.41], Standard Error of Mean 0.87

5. Secondary Outcome: Change From Treatment Baseline in SHAPS Total Score at Treatment Week 6 (fITT)
Description: as for outcome 4
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: The fITT analysis set included all enrolled participants who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-treatment baseline assessment of MADRS during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 77
scores on a scale | -3.7 (0.55) | -4.5 (0.55)
Statistical Analysis 1: Comparison: Double-blind Treatment + Withdrawal Period: Placebo vs Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg); Test type: Superiority; p = 0.2503, Mixed Models Analysis; Least Squares Mean Difference = -0.8, 80% CI 1-sided [upper limit 0.10], Standard Error of Mean 0.73

6. Secondary Outcome: Change From Treatment Baseline in Clinical Global Impression - Severity (CGI-S) Score at Treatment Week 6 (eITT Population)
Description: CGI-S provides an overall clinician-determined summary measure of severity of participant's illness that considers all available information, including knowledge of participant's history, psychosocial circumstances, symptoms, behavior, and impact of symptoms on participant's ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Participant is assessed on severity of mental illness at time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill participants. Negative change in score indicates improvement.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: eITT analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, had at least 1 post-baseline MADRS assessment during treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
Scores on a scale | -0.76 (0.858) [lower limit 0.858] | -0.92 (1.039) [lower limit 1.039]

7. Secondary Outcome: Change From Treatment Baseline in CGI-S Score at Treatment Week 6 (fITT Population)
Description: CGI-S provides an overall clinician-determined summary measure of severity of participants illness that considers all available information, including knowledge of participant's history, psychosocial circumstances, symptoms, behavior, and impact of symptoms on participant's ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Participant is assessed on severity of mental illness at time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill participants. Negative change in score indicates improvement.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: fITT analysis set included all enrolled participants who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-treatment baseline assessment of MADRS during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 77
Scores on a scale | -0.67 (0.880) | -0.87 (1.005)

8. Secondary Outcome: Change From Treatment Baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) Total Score at Treatment Week 6 (eITT Population)
Description: The SMDDS is a 16-item patient reported outcome (PRO) measure. Each item was rated by the participant according to a 5-point Likert scale. Participants respond to each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"). Before summing the items to create a total score, item 11 ("how often did you have a poor appetite") and item 12 ("how often did you over eat") were combined into a single score by selecting the highest severity on either item. The total score was then created by summing the responses on the 15 items. The total score ranged from 0 to 60. The SMDDS uses a 7-day recall period and verbal rating scales. Higher score indicates more severe depressive symptomatology. Negative change from baseline indicates improvement.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: The eITT analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
Scores on a scale | -8.49 (9.567) [lower limit 9.567] | -8.03 (9.957) [lower limit 9.957]

9. Secondary Outcome: Change From Treatment Baseline in SMDDS Total Score at Treatment Week 6 (fITT Population)
Description: as for outcome 8
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 80
Scores on a scale | -6.91 (9.996) | -8.16 (9.470)

10. Secondary Outcome: Number of Participants With Self-Assessment of Treatment Experience (SATE) Questionnaire at Treatment Week 6 (eITT Population)
Description: SATE questionnaire is a 3-item self-reported scale designed to provide additional information regarding participant's subjective experience while taking treatment. This was internal Janssen questionnaire and questions were asked to participant weekly by the Q1.6-app. For rating overall depression: participant selected one option out of Improved, not changed or got worse; for depression improvement: participant selected one option out of slightly improved, much improved or very much improved; and for depression worsen: participant selected slightly worse, much worse or very much worse.
Time Frame: Treatment Week 6
Population: The eITT analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'n' (number analyzed) refers to all participants evaluable for specified categories. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 40 | 30
Participants
  Overall Depression (Got worse) | 1 | 0
  Overall Depression (Not changed) | 12 | 9
  Overall Depression (Improved) | 27 | 21
  Depression Worsened (Slightly worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Slightly worse) | 1 |
  Depression Worsened (Much worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Much worse) | 0 |
  Depression Worsened (Very much worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Very much worse) | 0 |
  Depression Improvement (Slightly improved): number analyzed (Participants) | 27 | 21
  Depression Improvement (Slightly improved) | 13 | 15
  Depression Improvement (Much improved): number analyzed (Participants) | 27 | 21
  Depression Improvement (Much improved) | 11 | 6
  Depression Improvement (Very Much Improved): number analyzed (Participants) | 27 | 21
  Depression Improvement (Very Much Improved) | 3 | 0

11. Secondary Outcome: Number of Participants With SATE Questionnaire at Treatment Week 6 (fITT Population)
Description: as for outcome 10
Time Frame: Treatment Week 6
Population: (fITT) analysis set included all enrolled participants who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-treatment baseline assessment of MADRS during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure. Here 'n' (number analyzed) refers to all participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 49 | 42
Participants
  Overall Depression (Got worse) | 1 | 0
  Overall Depression (Not changed) | 15 | 12
  Overall Depression (Improved) | 33 | 30
  Depression Worsened (Slightly worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Slightly worse) | 1 |
  Depression Worsened (Much worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Much worse) | 0 |
  Depression Worsened (Very much worse): number analyzed (Participants) | 1 | 0
  Depression Worsened (Very much worse) | 0 |
  Depression Improvement (Slightly improved): number analyzed (Participants) | 33 | 30
  Depression Improvement (Slightly improved) | 18 | 20
  Depression Improvement (Much improved): number analyzed (Participants) | 33 | 30
  Depression Improvement (Much improved) | 12 | 9
  Depression Improvement (Very Much Improved): number analyzed (Participants) | 33 | 30
  Depression Improvement (Very Much Improved) | 3 | 1

12. Secondary Outcome: Change From Treatment Baseline in Hamilton Anxiety Scale 6 (HAM-A6) Total Score at Treatment Week 6 (eITT Population)
Description: HAM-A scale assesses severity of different anxiety-related symptoms with a score range of 0 to 52. Higher score indicated severity in anxiety symptoms. Each of the 14 items is rated by clinician on a 5-point scale ranging from 0 (not present) to 4 (maximum degree). HAM-A6 is a uni-dimensional, 6-item subscale derived from HAM-A. HAM-A6 comprises of five psychic anxiety symptoms: anxious mood, psychic tension, fears, intellectual disturbances, and anxious behaviour observed at the interview, as well as one somatic item, muscular tension. HAM-A6 subscale score ranges from 0 to 24, with higher scores indicating greater severity of core symptoms.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: eITT analysis set included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
scores on a scale | -2.19 (2.837) [lower limit 2.837] | -2.73 (2.651) [lower limit 2.651]

13. Secondary Outcome: Change From Treatment Baseline in HAM-A6 Total Score at Treatment Week 6 (fITT)
Description: as for outcome 12
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: (fITT) analysis set included all enrolled participants who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-treatment baseline assessment of MADRS during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 77
scores on a scale | -1.67 (2.842) | -2.68 (2.562)

14. Secondary Outcome: Change From Treatment Baseline in Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) Score at Treatment Week 6 (eITT Population)
Description: SIGH-A is a 14-item scale to measure severity of different anxiety-related symptoms in participants. Each of the 14 items is rated by the clinician on a 5-point scale ranging from 0 (not present) to 4 (maximum degree). The SIGH-A total score is calculated by summing the 14 item scores, and ranges from 0 to 56 where higher score indicates worsening.
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 59 | 59
scores on a scale | -5.37 (6.549) [lower limit 6.549] | -5.85 (5.369) [lower limit 5.369]

15. Secondary Outcome: Change From Treatment Baseline in SIGH-A Score at Treatment Week 6 (fITT Population)
Description: as for outcome 14
Time Frame: Treatment Baseline up to Week 6 of DB-treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 81 | 77
scores on a scale | -4.35 (6.193) | -5.47 (4.988)

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-67953964
Description: Cmax was defined as maximum observed plasma concentration of JNJ-67953964.
Time Frame: Week 1: Day 29, Week 3: Day 43, Week 6 (Day 64)
Population: eITT population included all enrolled lead-in placebo non-responders who were randomized into a treatment period, received at least 1 dose of study medication, and had at least 1 post-baseline MADRS assessment during the treatment period. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure. Here 'n' (number analyzed) refers to all participants evaluable for specified time point categories.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 58
nanograms per milliliter (ng/mL)
  Week 1 (Day 29) | 32.7 (10.9)
  Week 3 (Day 43) | 33.5 (11.1)
  Week 6 (Day 64): number analyzed (Participants) | 56
  Week 6 (Day 64) | 34.3 (11.1)

17. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 24 Hours Post-dose (AUC[0-24h]) of JNJ-67953964
Description: AUC(0-24h) was defined as the area under the plasma concentration-time curve from time of administration to 24 hours.
Time Frame: 0 to 24 hours Post dose on Week 1: Day 29, Week 3: Day 43, Week 6: Day 64
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 58
nanograms*hour per milliliter (ng*h/mL)
  Week 1 (Day 29) | 361 (156)
  Week 3 (Day 43) | 377 (164)
  Week 6 (Day 64): number analyzed (Participants) | 56
  Week 6 (Day 64) | 378 (163)

18. Secondary Outcome: Area Under Plasma Concentration-Time Curve at Steady State (AUCss) of JNJ-67953964
Description: AUCss was defined as the area under plasma concentration-time curve at Steady State (AUCss) of JNJ-67953964.
Time Frame: Week 1: Day 29, Week 3: Day 43, Week 6: Day 64
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 58
ng*h/mL
  Week 1 (Day 29) | 380 (151)
  Week 3 (Day 43) | 380 (151)
  Week 6 (Day 64): number analyzed (Participants) | 56
  Week 6 (Day 64) | 379 (153)

19. Secondary Outcome: Predose (Trough) Plasma Concentration (C0h) of JNJ-67953964
Description: C0h was defined as predose plasma Concentration of JNJ-67953964.
Time Frame: Predose on Week 1: Day 29, Week 3: Day 43, Week 6: Day 64
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
Number analyzed (Participants) | 58
nanograms per milliliter (ng/ml)
  Week 1 (Day 29) | 8.62 (4.27)
  Week 3 (Day 43) | 9.40 (4.69)
  Week 6 (Day 64): number analyzed (Participants) | 56
  Week 6 (Day 64) | 9.48 (4.83)

ADVERSE EVENTS:
Time Frame: Up to Week 11
Description: Full Safety analysis set included all enrolled participants who received at least 1 dose of study drug in treatment period.
Arm/Group | Lead in Period: Placebo | Double-blind Treatment + Withdrawal Period: Placebo | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/169 | 1/84 | 0/85
Other Adverse Events (participants affected / at risk) | 21/169 | 10/84 | 23/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead in Period: Placebo (N=169) | Double-blind Treatment + Withdrawal Period: Placebo (N=84) | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg) (N=85)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead in Period: Placebo (N=169) | Double-blind Treatment + Withdrawal Period: Placebo (N=84) | Double-blind Treatment + Withdrawal Period: JNJ-67953964 10 Milligrams (mg) (N=85)
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 7
Nasopharyngitis (Infections and infestations) | 6 | 3 | 6
Headache (Nervous system disorders) | 11 | 7 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03559192/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT03559192/SAP_001.pdf